CLINICAL TRIAL: NCT07236398
Title: Modified Left Atrial Maze Procedure: Achieving a Balance Between Safety and Efficacy in Concomitant Atrial Fibrillation Ablation
Brief Title: Modified Left Atrial Maze Procedure for Concomitant AF Ablation
Status: Enrolling by invitation | Type: Observational
Sponsor: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Myriam Addi, Principal Investigator, Department of Cardiovascular Surgery, University Hospital of Toulouse, University Paul Sabatier of Toulouse
Other Study IDs: UPaulSabatierToulouse1
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Cardiac Arrhythmia
Keywords: atrial fibrillation; surgical ablation; left Maze; cardiac surgery; rythm monitoring
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Modified left atrial Maze procedure performed concomitantly with cardiac surgery, including left atrial appendage closure, using bipolar radiofrequency and/or cryotherapy. — Patients undergo a standardized modified left atrial Maze procedure during cardiac surgery. The procedure includes pulmonary vein isolation using a BOX lesion set (bipolar radiofrequency clamp) for non-mitral surgeries, and an additional mitral line performed with cryotherapy for mitral valve surgeries. Left atrial appendage closure is systematically performed by excision-suture or AtriClip placement.
  Postoperative management includes beta-blockers, amiodarone when indicated, and lifelong anticoagulation according to guidelines. Rhythm evaluation is conducted at 3 and 12 months using ECG, 24-hour Holter monitoring, or pacemaker interrogation, along with quality-of-life assessment.

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia and affects up to 60% of patients undergoing cardiac surgery. Restoring sinus rhythm improves symptoms, reduces stroke risk, and prevents heart failure. Despite guideline recommendations, surgical ablation remains underused.

This study evaluates the safety and effectiveness of a standardized modified left atrial Maze procedure performed concomitantly with cardiac surgery and identifies early predictors of long-term rhythm success. The procedure consists of creating left atrial lesion sets using radiofrequency, cryothermy, or both, and systematically closing the left atrial appendage to reduce thromboembolic risk.

This prospective single-center observational study includes 151 patients undergoing concomitant AF ablation. Follow-up is performed at 3, 6, and 12 months with clinical evaluation, ECG, 24-hour Holter monitoring, pacemaker interrogation when applicable, and a standardized quality-of-life questionnaire.

The primary endpoint is sinus rhythm maintenance at 12 months. Secondary endpoints include operative mortality, neurological events, pacemaker implantation, reoperation for bleeding, and quality-of-life changes. The study aims to provide new insights into predictors of success and support standardized follow-up strategies for surgical AF ablation.

DETAILED DESCRIPTION:
This prospective observational registry was designed to evaluate the outcomes, safety profile, and predictive factors associated with a standardized modified left atrial Maze procedure performed concomitantly with cardiac surgery. The study focuses on the application of a reproducible lesion set, including a complete posterior left atrial "BOX" isolation and systematic left atrial appendage (LAA) closure, using bipolar radiofrequency, cryothermy, or a combination of both energy sources. The protocol reflects a structured institutional strategy developed at the University Hospital of Toulouse, allowing consistent perioperative management, uniform rhythm follow-up, and systematic quality-of-life assessment.

The modified left atrial Maze procedure aims to interrupt reentrant electrical circuits responsible for atrial fibrillation (AF) through the creation of continuous, transmural scar lines. In non-mitral procedures, the lesion set consists of pulmonary vein isolation and roof and floor lines creating a posterior "BOX." For mitral valve surgery, the standard lesion set is supplemented by a mitral isthmus line applied endocardially and epicardially to ensure transmurality. The LAA is excluded either through surgical excision with suture closure or via an external clip device. All lesion sets are performed concomitantly with the index cardiac procedure under cardiopulmonary bypass.

Postoperative management follows standardized institutional protocols including early beta-blockade, short-term amiodarone when indicated, rhythm monitoring, and systematic lifelong anticoagulation based on current guidelines. The structured follow-up schedule includes rhythm assessment by ECG, 24-hour Holter monitoring, or pacemaker interrogation at 3 and 12 months. Quality of life is assessed at baseline, 3 months, and 12 months using a simplified validated questionnaire derived from the SF-36 instrument.

Registry quality procedures include predefined data validation rules, routine checks for missing or inconsistent entries, and verification of collected data against source clinical records. All variables are defined within a standardized data dictionary specifying coding conventions, units, and clinically relevant thresholds. Data entry is performed by trained personnel within secured institutional electronic systems governed by the French MR-004 regulatory framework for clinical data handling. Periodic oversight is provided by the institutional data protection officer.

The sample size reflects the total number of eligible consecutive patients undergoing concomitant surgical AF ablation within the predefined inclusion period. Missing data are handled using a complete-case approach when the proportion of missing values remains below 5%, consistent with the predefined statistical plan. No imputation is performed when missingness is low and not expected to influence outcome distribution.

Statistical analyses include descriptive evaluation of the cohort, comparison of baseline characteristics according to sinus rhythm status at one year, and assessment of factors associated with rhythm outcomes. Quantitative variables are analyzed using non-parametric tests in the presence of non-normal distributions, and qualitative variables using chi-square methods. Univariate logistic regression identifies candidate variables associated with maintenance of sinus rhythm. Variables with p < 0.10 are entered into a multivariable logistic regression model using a backward elimination procedure. Analytical results are reported as odds ratios with 95% confidence intervals. All analyses follow predefined methodological standards and aim to identify early predictors of rhythm success following concomitant AF ablation.

This registry is intended to provide detailed and high-quality clinical data to support the evaluation of a standardized approach to surgical AF ablation, promote broader adoption of effective lesion sets, and inform future guideline development regarding perioperative rhythm management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Documented history of atrial fibrillation
* Scheduled for cardiac surgery
* Able to understand study information and provide non-opposition consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective single-center observational cohort includes adult patients with documented atrial fibrillation undergoing cardiac surgery at the University Hospital of Toulouse. All eligible patients during the inclusion period were consecutively enrolled and followed for one year.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Maintenance of sinus rhythm at 12 months after modified left atrial Maze procedure, assessed by 24-hour Holter monitoring or pacemaker interrogation | Sinus rhythm will be assessed at 12 months post-ablation using 24-hour Holter monitoring or pacemaker interrogation. Early rhythm assessment at 3 months is also performed for monitoring purposes.

CONTACTS AND LOCATIONS:
Locations (1):
- Myriam ADDI, Toulouse, French (France), France